CLINICAL TRIAL: NCT03897738
Title: Clinical Evaluation of Effectiveness and Safety of Combined Use of Dietary Supplements Amberen and Smart B in Women With Climacteric Syndrome in Perimenopause
Brief Title: Clinical Evaluation of Effectiveness and Safety of Amberen and Smart B in Perimenopausal Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Kuznetsova Irina, Chief Researcher, Scientific Research Centre, Women's Health Scientific Research Department, I.M. Sechenov First Moscow State Medical University, University hospital #2, Obstetrics and Gynecology clinic., I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AmberenSmartB-2019
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Perimenopause, Climacteric Syndrome
Keywords: succinate; B complex vitamins; perimenopause

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amberen and Smart B (Experimental): Amberen - a dietary supplement: 2 capsules (one while capsule 200 mg and one orange capsule 200 mg) are taken once a day with a meal, preferably after breakfast, for 3 months.
  SMART В - a dietary supplement: 1 capsule per day (166 mg) is taken once a day with a meal, preferably after breakfast, for 3 months, concurrently with Amberen.
  Interventions: Dietary Supplement: Amberen; Dietary Supplement: Smart B
- Placebo (Placebo Comparator): Placebo is taken as follows: 3 capsules (one while capsule 200 mg, one orange capsule 200 mg, one capsule 166mg) are taken once a day with a meal, preferably after breakfast, for 3 months.
  Placebo capsules are identical to Amberen and Smart B capsules.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Amberen — Amberen is a succinate-based dietary supplement previously shown to help provide relief for common menopausal symptoms.
  Arms: Amberen and Smart B
Dietary Supplement: Smart B — Smart B contains vitamins B1, B2, B6, B9, B12 and sodium fumarate.
  Arms: Amberen and Smart B
Dietary Supplement: Placebo — Placebo capsules are identical to Amberen and Smart B capsules.
  Arms: Placebo

SUMMARY:
To evaluate effectiveness and safety of combined use of dietary supplements Amberen and Smart B in women with a typical (without complications) form of climacteric syndrome, with mild to moderate symptoms in perimenopause.

DETAILED DESCRIPTION:
1. To evaluate effectiveness of combined use of dietary supplements Amberen and Smart B in women vasomotor, psychosomatic, psychological and other climacteric symptoms in perimenopause.
2. To evaluate safety of combined use of dietary supplements Amberen and Smart B in women with vasomotor, psychosomatic, psychological and other climacteric symptoms in perimenopause.
3. To develop recommendations for combined use of dietary supplements Amberen and Smart B for women with vasomotor, psychosomatic, psychological and other climacteric symptoms in perimenopause.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, 50 years of age or younger;

  * Subjects in the second phase of menopausal transition as per STRAW 10+ i.e. interval of amenorrhea 60 days or more (with regular menstrual cycle during earlier reproductive stages).
  * Subjects with diagnosis of mild to moderate climacteric syndrome;
  * Recent (up to 12 months prior to study enrollment) breast exam results, including mammogram, that rule out malignancies;
  * Recent (up to 3 years prior to study enrollment) cytological screening that rules out vaginal cervix malignancies.
  * Ability to read and understand informed consent form for the study's participation;
  * Ability to adhere to the conditions of the study.

Exclusion Criteria:

* • Postmenopause, including surgical menopause.

  * Presence of hormone-dependent cancers;
  * Presence of other cancers, not in full remission with no recurrence for 5 years or more;
  * Planned hospitalization in the next 6 months;
  * Presence of hormonally-active extragenital endocrine diseases (diabetes; diseases of thyroid, adrenal, pituitary) that require prolonged or life-long therapies
  * Surgical interventions on sex organs or breasts, 1 year or less prior to the screening;
  * Gynecological conditions that may require hormonal therapies or surgeries (uterine myoma, endometriosis, endometrial hyperplasia etc.);
  * Currently undergoing or planning to utilize assisted reproductive technologies;
  * Any abdominal surgeries within less than 3 months prior to the screening;
  * HRT including MHRT or hormonal contraceptives - current or within less than 3 months prior to the screening;
  * Psychiatric conditions;
  * Patients taking any other dietary supplements that can affect climacteric syndrome within the last month before enrolling in the trial;
  * High risk of non-compliance.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
"Heart beating quickly and strongly" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 1 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Feeling tense or nervous" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 2 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Difficulty sleeping" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 3 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Increased Excitability" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 4 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Panic attacks" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 5 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Difficulty concentrating" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 6 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Feeling tired or lacking energy" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 7 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Loss of interest in most things" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 8 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Feeling of sadness or depression" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 9 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Crying spells" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 10 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Irritability" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 11 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Feeling dizzy or faint" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 12 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Pressure or tightness in head or body" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 13 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Parts of body feeling numb or tingling" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 14 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Headaches" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 15 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Muscle or joint pains" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 16 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Loss of feeling in hands or feet" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 17 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Breathing difficulties" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 18 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Hot flushes" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 19 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Night sweats" symptom (Greene Climacteric Scale) | 90 days and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 20 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
"Loss of interest in sex" symptom (Greene Climacteric Scale) | 90 and 180 days
  Statistically significant change in designated symptom severity, compared between arms. This is question 21 of the Greene Climacteric Scale; the subjects rank degrees of bother of the symptom as 1 = "not at all"; 2 = "a little bit"; 3 = "quite a bit"; 4 = "extremely"
Blood plasma estradiol levels, pg/ml | 90 and 180 days
  Statistically significant changes in the levels, compared between arms

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (State anxiety sub-scale) | 90 and 180 days
  Statistically significant change of the score in corresponding sub-scale. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
State-Trait Anxiety Inventory (Trait anxiety sub-scale) | 90 and 180 days
  Statistically significant change of the score in corresponding sub-scale. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
State-Trait Anxiety Inventory (Actual anxiety, combination of state and trait sub-scales ) | 90 and 180 days
  Statistically significant change of the score in corresponding sub-scale. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Well-being sub-score (Russian well-being, activity and mood questionnaire) | 90 and 180 days
  Statistically significant change in designated symptom severity, compared between arms. The sub-scale score varies from 10 to 70 points, with the higher score corresponding to more positive self-evaluation of well-being.
Activity sub-score (Russian well-being, activity and mood questionnaire) | 90 and 180 days
  Statistically significant change in designated symptom severity, compared between arms. The sub-scale score varies from 10 to 70 points, with the higher score corresponding to more positive self-evaluation of one's activity.
Mood sub-score (Russian well-being, activity and mood questionnaire) | 90 and 180 days
  Statistically significant change in designated symptom severity, compared between arms. The sub-scale score varies from 10 to 70 points, with the higher score corresponding to more positive self-evaluation of one's mood.
Anxiety sub-score (measured by Hospital Anxiety and Depression Scale) | 90 and 180 days
  Statistically significant change in designated symptom severity, compared between arms. The scores range from 0 to 21.
  0-7 = Normal 8-10 = Borderline abnormal 11-21 = Abnormal
Depression sub-score (measured by Hospital Anxiety and Depression Scale) | 90 and 180 days
  Statistically significant change in designated symptom severity, compared between arms. The scores range from 0 to 21.
  0-7 = Normal 8-10 = Borderline abnormal 11-21 = Abnormal

CONTACTS AND LOCATIONS:
Locations (1):
- Sechenov First Moscow Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kachko VA, Shulman LP, Kuznetsova IV, Uspenskaya YB, Burchakov DI. Clinical Evaluation of Effectiveness and Safety of Combined Use of Dietary Supplements Amberen(R) and Smart B(R) in Women with Climacteric Syndrome in Perimenopause. Adv Ther. 2024 Aug;41(8):3183-3195. doi: 10.1007/s12325-024-02910-0. Epub 2024 Jun 21. PMID 38904899